CLINICAL TRIAL: NCT04841382
Title: Physician Assessment of the Clinical Utility of a Patient-Specific 3D Electro-Anatomical Heart Model in VT Ablation
Acronym: ACE-VT
Status: Terminated | Type: Observational
Why Stopped: Sponsor
Sponsor: CardioSolv Ablation Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: REDD-0018
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Monomorphic Ventricular Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Supporting information. — CardioSolv Software System is a software-based medical device meant which creates a patient-specific 3D heart model that provides physiologic information.

SUMMARY:
ACE-VT is a clinical pilot study designed to evaluate the ability of the CardioSolv Software System to generate an output for the physician to review in a timely fashion, consistent with the standard of care VT ablation workflow. This study will assess the acute effectiveness of using the CardioSolv Software System output as additional supporting information during ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant meets standard criteria for VT ablation and is scheduled for VT ablation by their cardiologist or electrophysiologist
2. 18 to 85 years of age
3. VT and ischemic cardiomyopathy
4. A pre-procedure MRI with LGE is available (performed within 1 year of procedure, unless an MI has occurred since MRI) with adequate image for analysis
5. Participant is able and willing to provide written informed consent

Exclusion Criteria:

1. Contradiction to MRI (except those with MRI compatible pacemaker/ICD/CRT devices implanted or site has approved procedure for MRI of non-compatible devices).
2. Participant implanted with an LVAD.
3. Enrolled in another non-imaging intervention assignment study that could confound the results of this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with monomorphic VT secondary to ischemic cardiomyopathy scheduled for a VT ablation procedure will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Time to Receipt of 3D Heart Model | 24 hours
  Verify that the CardioSolv Software System is able to receive and process input data and generate the expected output available for viewing by the physician in less than 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Saman Nazarian, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Upenn, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided